CLINICAL TRIAL: NCT00825565
Title: Open-label, Pilot Study to Investigate the Safety and Tolerability of Alwextin 3.0% Cream in the Treatment of Epidermolysis Bullosa
Brief Title: Study of Alwextin® Cream in Treating Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Amy Paller, Professor and Chair of Deparment of Dermatology, Professor of Pediatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alwextin 3.0%-04
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Epidermolysis Bullosa
Keywords: Epidermolysis bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Allantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alwextin cream (Experimental): 8 subjects enrolled in this single study arm. All 8 subjects completed the study.
  Interventions: Drug: Alwextin cream

INTERVENTIONS:
Drug: Alwextin cream — Alwextin cream contains active ingredient, allantoin 3%. Use 1 application daily for 3 month duration.
  Other Names: Alwextin; Alwyn; allantoin

SUMMARY:
The purpose of this study is to determine how safe and effective allantoin 3% cream (Alwextin) is in improving the healing of recurrent skin lesions and reducing overall blistering in people with epidermolysis bullosa (EB). Allantoin 3% cream is applied topically to the entire body once daily.

DETAILED DESCRIPTION:
Potential subjects came to the for a screening visit. Eligible subjects had baseline assessments performed and were provided study medication, allantoin 3% cream. Subjects were instructed to apply the study medication to the entire body once daily and to keep daily record of study medication use. Subjects returned every 4 weeks for a total of 12 weeks for repeat assessments.

ELIGIBILITY:
Inclusion Criteria:

* history of epidermolysis bullosa

Exclusion Criteria:

* use of any skin product containing allantoin for 30 days prior to enrollment

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Robert and Ann Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were identified at regularly scheduled clinic visits with the Principal Investigator at Children's Memorial Hospital.
Pre-assignment Details: Subjects were instructed to discontinue use of allantoin 1.5% cream (Alwyn) for at least 30 days prior to initiating the study medication, allantoin 3% cream (Alwextin).
Groups:
- Allantoin 3% Cream: This is an open-label study in which all enrolled subjects were assigned to receive the study medication, allantoin 3% cream. Subjects were required to have a diagnosis of Epidermolysis Bullosa (EB). The diagnosis of EB was based on diagnostic immunomapping, electron microscopy, or the principal investigator's judgment based on clear clinical characteristics. Subjects were instructed to apply allantoin 3% cream once daily to the entire body.
Period: Overall Study
Arm/Group | Allantoin 3% Cream
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allantoin 3% Cream
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Blister/Erosion Reduction Based on Change in Body Surface Area (BSA) Coverage
Description: A common measure of the degree of involvement in skin disease is the Body Surface Area Index (BSAI). This measure is also commonly used in psoriasis studies. It is a global measure of disease "spread" with weighting factors.
Time Frame: baseline and then every 4 weeks for a total of 12 weeks
Population: Subjects who used allantoin 3% cream for an entire month prior to the BSA monthly assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of BSA involvement
Groups:
- Allantoin 3% Cream: Subjects were instructed to apply allantoin 3% cream once daily to the entire body.
Arm/Group | Allantoin 3% Cream
Number analyzed (Participants) | 8
percentage of BSA involvement
  Baseline assessment | 57.25 (19.1)
  Week 4 assessment | 39.40 (24.1)
  Week 8 assessment | 27.25 (17.9)
  Week 12 assessment | 25.45 (21.1)

2. Primary Outcome: Target Wound Size Reduction or Closure
Description: EB patients may have chronic wounds which are resistant to healing. Wound size may be very large and the probability of total wound closure with currently available treatments is unlikely. Reduction in the size of wounds may be clinically important to the rate of infection and pain. If a patient has a reduction in the size of wounds which are refractory to healing, this may be seen as a positive outcome. Wound size reduction is one of the primary assessments used to determine the efficacy of the study cream.
  Wounds which had been present for at least several weeks prior to study entry were measured by using VISITRAK Digital, a Smith and Nephew wound tracing and measurement system that will calculate the length and width of the lesion (class 1 medical device; FDA listing designation E142354FDA). Only one target lesion per patient was used for the study assessment. At each subsequent study until the final visit, the target lesion was evaluated using VISITRAK Digital.
Time Frame: baseline and then every 4 weeks for a total of 12 weeks
Population: Subjects who used allantoin 3% cream on the target wound daily up to full closure of that wound were included in the analysis.
Measure: Number; unit: number of unhealed target wounds
Groups:
- Allantoin 3% Cream: Subjects were instructed to apply allantoin 3% cream once daily to the target lesion area for assessing the impact on target wound closure.
Arm/Group | Allantoin 3% Cream
Number analyzed (Participants) | 8
number of unhealed target wounds
  Baseline assessment | 8
  Week 12 assessment | 1

3. Primary Outcome: Physician Global Assessment of Severity (PGAS)
Description: The FDA has suggested that a global measure of severity might be the best way to assess EB from visit to visit. Assessment score may be influenced by other clinical observations in addition to the percentage of body affected by blistering and erosions. The assessment was intended to be a "global impression."
  This scale produced a score with the following correlations:
  0 = clear (no blistering/erosions) 1-2 = almost clear (infrequent blistering and erosions) 3-4 = mild disease (up to 15% of body affected) 5-6 = moderate disease (between 16-25% of body affected) 7-8 = severe disease (between 26-50% of body affected) 9-10 = very severe disease (greater than 50% of body affected)
Time Frame: baseline and then every 4 weeks for a total of 12 weeks
Population: One subject discontinued after week 3. One subject discontinued at Month 2. Only data presented for subjects who used cream on entire body for the entire month was used in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Alwextin Cream
Number analyzed (Participants) | 8
Participants
  Baseline: PGAS score of 1 | 0
  Baseline: PGAS score of 2 | 0
  Baseline: PGAS score of 3 | 0
  Baseline: PGAS score of 4 | 0
  Baseline: PGAS score of 5 | 0
  Baseline: PGAS score of 6 | 0
  Baseline: PGAS score of 7 | 1
  Baseline: PGAS score of 8 | 2
  Baseline: PGAS score of 9 | 3
  Baseline: PGAS score of 10 | 2
  Month 1: number analyzed (Participants) | 7
  Month 1: PGAS score of 1 | 0
  Month 1: PGAS score of 2 | 0
  Month 1: PGAS score of 3 | 0
  Month 1: PGAS score of 4 | 0
  Month 1: PGAS score of 5 | 2
  Month 1: PGAS score of 6 | 1
  Month 1: PGAS score of 7 | 2
  Month 1: PGAS score of 8 | 1
  Month 1: PGAS score of 9 | 0
  Month 1: PGAS score of 10 | 1
  Month 2: number analyzed (Participants) | 6
  Month 2: PGAS score of 1 | 0
  Month 2: PGAS score of 2 | 0
  Month 2: PGAS score of 3 | 0
  Month 2: PGAS score of 4 | 1
  Month 2: PGAS score of 5 | 2
  Month 2: PGAS score of 6 | 1
  Month 2: PGAS score of 7 | 1
  Month 2: PGAS score of 8 | 0
  Month 2: PGAS score of 9 | 1
  Month 2: PGAS score of 10 | 0
  Month 3: number analyzed (Participants) | 4
  Month 3: PGAS score of 1 | 0
  Month 3: PGAS score of 2 | 0
  Month 3: PGAS score of 3 | 0
  Month 3: PGAS score of 4 | 2
  Month 3: PGAS score of 5 | 0
  Month 3: PGAS score of 6 | 0
  Month 3: PGAS score of 7 | 1
  Month 3: PGAS score of 8 | 0
  Month 3: PGAS score of 9 | 1
  Month 3: PGAS score of 10 | 0

4. Primary Outcome: Physician Assessment of Individual Signs
Description: In addition to skin blistering and erosions, people with EB experience other symptoms, such as erythema on unblistered skin, wound oozing, weeping, and crusting. These symptoms may vary with area of the body evaluated.
  This scale evaluates the following signs: Blistering and erosions, oozing/weeping/crusting, pruritis, erythema on unblistered surrounding skin, pain, milia Each of these signs will be scored in 4 body areas: head/neck, upper limbs, trunk, lower limbs The following scale is used:0 = clear 1 = almost clear 2 = mild 3 = moderate 4 = severe
Time Frame: baseline and at 12 weeks
Population: Subjects who used cream on entire body for the entire month was used in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Head/Neck | Upper Limbs | Trunk | Lower Limbs
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  Pain-Baseline: Clear | 1 | 0 | 0 | 0
  Pain-Baseline: Almost Clear | 4 | 4 | 3 | 1
  Pain-Baseline: Mild | 2 | 1 | 0 | 1
  Pain-Baseline: Moderate | 0 | 1 | 3 | 2
  Pain-Baseline: Severe | 1 | 2 | 2 | 4
  Pain-Month 3: number analyzed (Participants) | 4 | 4 | 4 | 4
  Pain-Month 3: Clear | 2 | 2 | 2 | 2
  Pain-Month 3: Almost Clear | 0 | 0 | 0 | 0
  Pain-Month 3: Mild | 2 | 1 | 1 | 1
  Pain-Month 3: Moderate | 0 | 1 | 0 | 0
  Pain-Month 3: Severe | 0 | 0 | 1 | 1
  Pruritis-Baseline: Clear | 2 | 0 | 0 | 0
  Pruritis-Baseline: Almost Clear | 5 | 5 | 3 | 3
  Pruritis-Baseline: Mild | 1 | 0 | 0 | 2
  Pruritis-Baseline: Moderate | 0 | 0 | 2 | 2
  Pruritis-Baseline: Severe | 0 | 3 | 3 | 1
  Pruritus-Month 3: number analyzed (Participants) | 4 | 4 | 4 | 4
  Pruritus-Month 3: Clear | 3 | 2 | 2 | 2
  Pruritus-Month 3: Almost Clear | 0 | 1 | 1 | 1
  Pruritus-Month 3: Mild | 0 | 0 | 0 | 0
  Pruritus-Month 3: Moderate | 1 | 1 | 1 | 1
  Pruritus-Month 3: Severe | 0 | 0 | 0 | 0
  Blisters/Erosions-Baseline: Clear | 1 | 0 | 0 | 0
  Blisters/Erosions-Baseline: Almost Clear | 1 | 1 | 0 | 0
  Blisters/Erosions-Baseline: Mild | 4 | 1 | 2 | 0
  Blisters/Erosions-Baseline: Moderate | 2 | 4 | 3 | 3
  Blisters/Erosions-Baseline: Severe | 0 | 2 | 3 | 5
  Blisters/Erosions- Month 3: number analyzed (Participants) | 4 | 4 | 4 | 4
  Blisters/Erosions- Month 3: Clear | 0 | 0 | 0 | 0
  Blisters/Erosions- Month 3: Almost Clear | 2 | 0 | 1 | 1
  Blisters/Erosions- Month 3: Mild | 2 | 2 | 2 | 1
  Blisters/Erosions- Month 3: Moderate | 0 | 2 | 0 | 1
  Blisters/Erosions- Month 3: Severe | 0 | 0 | 1 | 1
  Oozing/Weeping/Crusting-Baseline: Clear | 1 | 0 | 0 | 0
  Oozing/Weeping/Crusting-Baseline: Almost Clear | 3 | 2 | 1 | 1
  Oozing/Weeping/Crusting-Baseline: Mild | 1 | 0 | 1 | 0
  Oozing/Weeping/Crusting-Baseline: Moderate | 3 | 5 | 3 | 3
  Oozing/Weeping/Crusting-Baseline: Severe | 0 | 1 | 3 | 4
  Oozing/Weeping/Crusting- Month 3: number analyzed (Participants) | 4 | 4 | 4 | 4
  Oozing/Weeping/Crusting- Month 3: Clear | 1 | 0 | 0 | 0
  Oozing/Weeping/Crusting- Month 3: Almost Clear | 1 | 1 | 2 | 1
  Oozing/Weeping/Crusting- Month 3: Mild | 0 | 1 | 1 | 1
  Oozing/Weeping/Crusting- Month 3: Moderate | 2 | 2 | 0 | 1
  Oozing/Weeping/Crusting- Month 3: Severe | 0 | 0 | 1 | 1
  Erythema-Baseline: Clear | 0 | 0 | 0 | 0
  Erythema-Baseline: Almost Clear | 3 | 2 | 1 | 0
  Erythema-Baseline: Mild | 4 | 1 | 1 | 3
  Erythema-Baseline: Moderate | 0 | 3 | 2 | 2
  Erythema-Baseline: Severe | 1 | 2 | 4 | 3
  Erythema- Month 3: number analyzed (Participants) | 4 | 4 | 4 | 4
  Erythema- Month 3: Clear | 1 | 1 | 1 | 1
  Erythema- Month 3: Almost Clear | 2 | 2 | 2 | 2
  Erythema- Month 3: Mild | 1 | 1 | 0 | 0
  Erythema- Month 3: Moderate | 0 | 0 | 1 | 1
  Erythema- Month 3: Severe | 0 | 0 | 0 | 0
  Milia-Baseline: Clear | 7 | 8 | 8 | 8
  Milia-Baseline: Almost Clear | 1 | 0 | 0 | 0
  Milia-Baseline: Mild | 0 | 0 | 0 | 0
  Milia-Baseline: Moderate | 0 | 0 | 0 | 0
  Milia-Baseline: Severe | 0 | 0 | 0 | 0
  Milia- Month 3: number analyzed (Participants) | 4 | 4 | 4 | 4
  Milia- Month 3: Clear | 3 | 3 | 3 | 4
  Milia- Month 3: Almost Clear | 1 | 0 | 1 | 0
  Milia- Month 3: Mild | 0 | 1 | 0 | 0
  Milia- Month 3: Moderate | 0 | 0 | 0 | 0
  Milia- Month 3: Severe | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For 12 week duration of study. Adverse events (AE) and serious adverse events (SAE_that were unresolved by study completion date were followed for an additional 1 month post-study completion.
Description: AE is defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical treatment or procedure. SAE meets any of these criteria: causes death, hospitalization, disability, or birth defect, is life-threatening, is an important medical event that may require intervention to prevent these outcomes.
Arm/Group | Allantoin 3% Cream
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allantoin 3% Cream (N=8)
red, itchy skin (Skin and subcutaneous tissue disorders) | 1 (1) — unlikely to be related to study medication
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — unlikely to be related to study medication
fever (General disorders) | 2 (2) — unlikely to be related to study medication
red spots on right foot (Skin and subcutaneous tissue disorders) | 1 (1) — unlikely to be related to study medication
red spots on left foot (Skin and subcutaneous tissue disorders) | 1 (1) — unlikely to be related to study medication
diarrhea (Gastrointestinal disorders) | 1 (1) — unlikely to be related to study medication
hematemesis (Gastrointestinal disorders) | 1 (1) — not related to study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No